CLINICAL TRIAL: NCT05096312
Title: A Randomized, Double Blind, Placebo-Controlled Clinical Trial of the Effects of Oral Zinc Gluconate Among Diagnosed Acne Vulgaris Patients
Brief Title: Effects of Oral Zinc Gluconate Among Acne Vulgaris Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Avenue Medical Center, Philippines (Other Government)
Responsible Party: Principal Investigator, Monique Lianne C. Lim-Ang, MD, MBA, DPDS, Principal Investigator, East Avenue Medical Center, Philippines
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAMC IERB 2018-52
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; zinc gluconate; inflammation; adapalene; benzoyl peroxide; Global Acne Grading System
MeSH Terms: conditions — Acne Vulgaris; Inflammation | interventions — gluconic acid; Adapalene; Benzoyl Peroxide; Gels; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zinc gluconate group (Active Comparator): interventions: Zinc gluconate (200g/capsule) one capsule once in the morning after breakfast for 60 days.
  Adapalene 0.3% + benzoyl peroxide 2.5% gel to be applied once at night for 60 days.
  Interventions: Dietary Supplement: Zinc gluconate; Drug: Adapalene 0.003 MG/MG / Benzoyl Peroxide 0.025 MG/MG Topical Gel [Epiduo]
- Placebo group (Placebo Comparator): interventions: Placebo capsule, one capsule once in the morning after breakfast for 60 days. Adapalene 0.3% + benzoyl peroxide 2.5% gel to be applied once at night for 60 days.
  Interventions: Drug: Adapalene 0.003 MG/MG / Benzoyl Peroxide 0.025 MG/MG Topical Gel [Epiduo]; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — oral zinc gluconate 200mg
  Other Names: Solgar zinc gluconate
  Arms: Zinc gluconate group
Drug: Adapalene 0.003 MG/MG / Benzoyl Peroxide 0.025 MG/MG Topical Gel [Epiduo] — Adapalene 0.3% + Benzoyl peroxide 2.5% gel applied once daily in the evening
  Other Names: Epiduo Forte
Other: Placebo — contains cornstarch
  Arms: Placebo group

SUMMARY:
Acne Vulgaris is one of the most common dermatologic diagnoses requiring long-term maintenance therapy. Promising results of oral zinc gluconate in improving acne vulgaris has been described.

A randomized, double blind, placebo-controlled clinical trial was utilized for this study with the objective to assess the efficacy of oral zinc gluconate in the improvement of disease activity in acne vulgaris patients as measured by the inflammatory score and Global Acne Grading System (GAGS) score.

DETAILED DESCRIPTION:
Acne has four main pathogenic contributors: follicular hyperkeratinization, increased sebum production, Propionibacterium acnes (P. acnes) within the follicle, and inflammation. Treatment options for acne vulgaris include benzoyl peroxide, topical and oral retinoids, topical and oral antimicrobials, oral corticosteroids, and physical modalities such as acne surgery, laser and light therapy. Reports show that antibiotic resistance is a growing issue in the treatment regimen of acne vulgaris, making it less and less suitable for long-term treatment, hence other options that can be substitutes or adjuncts to treatment may be useful in this condition. For long-term or maintenance therapy, physicians should consider effectivity, cost, and adverse effects. Several studies have explored the effect of oral zinc on acne vulgaris. Since zinc is more cost-effective and has less adverse effects compared to most antibiotics, this may prove helpful for the Filipino patient in terms of safety and economy for long-term therapy.

The aim of this study is to assess the efficacy of oral zinc gluconate in the improvement of disease activity in acne vulgaris patients, to determine the demographic and clinical profile of Acne Vulgaris patients, to determine the disease activity measured by the inflammatory score and GAGS score of acne vulgaris patients on initial consult, at 4 weeks, and at 8 weeks, and to determine if there is a significant difference in disease activity as measured by the inflammatory score and GAGS score among acne vulgaris patients given placebo and oral zinc gluconate.

A randomized, double blind, placebo-controlled clinical trial was utilized. Adults with moderate to severe acne vulgaris were included in the study. Patients were evaluated using the inflammatory score and Global Acne Grading System (GAGS) at the start, at midpoint, and at the end of the trial. One group of participants received zinc gluconate supplementation and another group received placebo for 60 days. All participants received topical adapalene 0.3% + Benzoyl peroxide 2.5% gel applied once daily in the evening. Improvement in acne severity was then determined and compared.

ELIGIBILITY:
Inclusion Criteria:

* Filipino patients, aged 18-27 years old
* New patients diagnosed with Acne Vulgaris with a Global Acne Grading System score of at least 19
* Able to read and write in English or Tagalog
* Seen at the Dermatology out-patient clinic of East Avenue Medical Center

Exclusion Criteria:

* Patients with other chronic dermatoses or systemic disease
* Taking oral supplements or medications within the past 4 weeks
* Patients who are pregnant or lactating

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Lianne C. Lim-Ang, MD,MBA,DPDS, Principal Investigator — East Avenue Medical Center
Locations (1):
- East Avenue Medical Center, Quezon City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhate K, Williams HC. Epidemiology of acne vulgaris. Br J Dermatol. 2013 Mar;168(3):474-85. doi: 10.1111/bjd.12149. PMID 23210645
- [Background] Humphrey S. Antibiotic resistance in acne treatment. Skin Therapy Lett. 2012 Oct;17(9):1-3. PMID 23032935
- [Background] Tan JK, Bhate K. A global perspective on the epidemiology of acne. Br J Dermatol. 2015 Jul;172 Suppl 1:3-12. doi: 10.1111/bjd.13462. PMID 25597339
- [Background] Collier CN, Harper JC, Cafardi JA, Cantrell WC, Wang W, Foster KW, Elewski BE. The prevalence of acne in adults 20 years and older. J Am Acad Dermatol. 2008 Jan;58(1):56-9. doi: 10.1016/j.jaad.2007.06.045. Epub 2007 Oct 22. PMID 17945383
- [Background] Goulden V, Stables GI, Cunliffe WJ. Prevalence of facial acne in adults. J Am Acad Dermatol. 1999 Oct;41(4):577-80. PMID 10495379
- [Background] Thiboutot DM, Dreno B, Abanmi A, Alexis AF, Araviiskaia E, Barona Cabal MI, Bettoli V, Casintahan F, Chow S, da Costa A, El Ouazzani T, Goh CL, Gollnick HPM, Gomez M, Hayashi N, Herane MI, Honeyman J, Kang S, Kemeny L, Kubba R, Lambert J, Layton AM, Leyden JJ, Lopez-Estebaranz JL, Noppakun N, Ochsendorf F, Oprica C, Orozco B, Perez M, Piquero-Martin J, See JA, Suh DH, Tan J, Lozada VT, Troielli P, Xiang LF. Practical management of acne for clinicians: An international consensus from the Global Alliance to Improve Outcomes in Acne. J Am Acad Dermatol. 2018 Feb;78(2 Suppl 1):S1-S23.e1. doi: 10.1016/j.jaad.2017.09.078. Epub 2017 Nov 8. PMID 29127053
- [Background] Stein Gold L, Weiss J, Rueda MJ, Liu H, Tanghetti E. Moderate and Severe Inflammatory Acne Vulgaris Effectively Treated with Single-Agent Therapy by a New Fixed-Dose Combination Adapalene 0.3 %/Benzoyl Peroxide 2.5 % Gel: A Randomized, Double-Blind, Parallel-Group, Controlled Study. Am J Clin Dermatol. 2016 Jun;17(3):293-303. doi: 10.1007/s40257-016-0178-4. PMID 26945741
- [Background] Al-Shobaili HA. Oxidants and anti-oxidants status in acne vulgaris patients with varying severity. Ann Clin Lab Sci. 2014 Spring;44(2):202-7. PMID 24795060
- [Background] Bray TM, Bettger WJ. The physiological role of zinc as an antioxidant. Free Radic Biol Med. 1990;8(3):281-91. doi: 10.1016/0891-5849(90)90076-u. PMID 2187766
- [Background] Prasad AS. Zinc is an Antioxidant and Anti-Inflammatory Agent: Its Role in Human Health. Front Nutr. 2014 Sep 1;1:14. doi: 10.3389/fnut.2014.00014. eCollection 2014. PMID 25988117
- [Background] Rostan EF, DeBuys HV, Madey DL, Pinnell SR. Evidence supporting zinc as an important antioxidant for skin. Int J Dermatol. 2002 Sep;41(9):606-11. doi: 10.1046/j.1365-4362.2002.01567.x. PMID 12358835
- [Background] Sardana K, Chugh S, Garg VK. The role of zinc in acne and prevention of resistance: have we missed the "base" effect? Int J Dermatol. 2014 Jan;53(1):125-7. doi: 10.1111/ijd.12264. No abstract available. PMID 24350859
- [Background] Buxaderas SC, Farre-Rovira R. Whole blood and serum zinc levels in relation to sex and age. Rev Esp Fisiol. 1985 Dec;41(4):463-70. PMID 4095368
- [Background] Amer M, Bahgat MR, Tosson Z, Abdel Mowla MY, Amer K. Serum zinc in acne vulgaris. Int J Dermatol. 1982 Oct;21(8):481-4. doi: 10.1111/j.1365-4362.1982.tb03188.x. PMID 6217164
- [Background] Arora PN, Dhillon KS, Rajan SR, Sayal SK, Das AL. Serum Zinc Levels in Cutaneous Disorders. Med J Armed Forces India. 2002 Oct;58(4):304-6. doi: 10.1016/S0377-1237(02)80083-1. Epub 2011 Jul 21. PMID 27407419
- [Background] Rostami Mogaddam M, Safavi Ardabili N, Maleki N, Soflaee M. Correlation between the severity and type of acne lesions with serum zinc levels in patients with acne vulgaris. Biomed Res Int. 2014;2014:474108. doi: 10.1155/2014/474108. Epub 2014 Jul 24. PMID 25157359
- [Background] Michaelsson G, Vahlquist A, Juhlin L. Serum zinc and retinol-binding protein in acne. Br J Dermatol. 1977 Mar;96(3):283-6. doi: 10.1111/j.1365-2133.1977.tb06138.x. PMID 139912
- [Background] Ozuguz P, Dogruk Kacar S, Ekiz O, Takci Z, Balta I, Kalkan G. Evaluation of serum vitamins A and E and zinc levels according to the severity of acne vulgaris. Cutan Ocul Toxicol. 2014 Jun;33(2):99-102. doi: 10.3109/15569527.2013.808656. Epub 2013 Jul 5. PMID 23826827
- [Background] Gupta M, Mahajan VK, Mehta KS, Chauhan PS. Zinc therapy in dermatology: a review. Dermatol Res Pract. 2014;2014:709152. doi: 10.1155/2014/709152. Epub 2014 Jul 10. PMID 25120566
- [Background] Bae YS, Hill ND, Bibi Y, Dreiher J, Cohen AD. Innovative uses for zinc in dermatology. Dermatol Clin. 2010 Jul;28(3):587-97. doi: 10.1016/j.det.2010.03.006. PMID 20510767
- [Background] Bibi Nitzan Y, Cohen AD. Zinc in skin pathology and care. J Dermatolog Treat. 2006;17(4):205-10. doi: 10.1080/09546630600791434. PMID 16971312
- [Background] Michaelsson G, Juhlin L, Ljunghall K. A double-blind study of the effect of zinc and oxytetracycline in acne vulgaris. Br J Dermatol. 1977 Nov;97(5):561-6. doi: 10.1111/j.1365-2133.1977.tb14136.x. PMID 145237
- [Background] Dreno B, Moyse D, Alirezai M, Amblard P, Auffret N, Beylot C, Bodokh I, Chivot M, Daniel F, Humbert P, Meynadier J, Poli F; Acne Research and Study Group. Multicenter randomized comparative double-blind controlled clinical trial of the safety and efficacy of zinc gluconate versus minocycline hydrochloride in the treatment of inflammatory acne vulgaris. Dermatology. 2001;203(2):135-40. doi: 10.1159/000051728. PMID 11586012
- [Background] Cunliffe WJ, Burke B, Dodman B, Gould DJ. A double-blind trial of a zinc sulphate/citrate complex and tetracycline in the treatment of acne vulgaris. Br J Dermatol. 1979 Sep;101(3):321-5. doi: 10.1111/j.1365-2133.1979.tb05626.x. PMID 159714
- [Background] Dreno B, Amblard P, Agache P, Sirot S, Litoux P. Low doses of zinc gluconate for inflammatory acne. Acta Derm Venereol. 1989;69(6):541-3. PMID 2575335
- [Background] Hillstrom L, Pettersson L, Hellbe L, Kjellin A, Leczinsky CG, Nordwall C. Comparison of oral treatment with zinc sulphate and placebo in acne vulgaris. Br J Dermatol. 1977 Dec;97(6):681-4. doi: 10.1111/j.1365-2133.1977.tb14277.x. PMID 146511
- [Background] Goransson K, Liden S, Odsell L. Oral zinc in acne vulgaris: a clinical and methodological study. Acta Derm Venereol. 1978;58(5):443-8. PMID 82356
- [Background] Verma KC, Saini AS, Dhamija SK. Oral zinc sulphate therapy in acne vulgaris: a double-blind trial. Acta Derm Venereol. 1980;60(4):337-40. doi: 10.2340/0001555560337340. PMID 6163281
- [Background] Sardana K, Garg VK. An observational study of methionine-bound zinc with antioxidants for mild to moderate acne vulgaris. Dermatol Ther. 2010 Jul-Aug;23(4):411-8. doi: 10.1111/j.1529-8019.2010.01342.x. PMID 20666829
- [Background] Vahlquist A, Michaelsson G, Juhlin L. Acne treatment with oral zinc and vitamin A: effects on the serum levels of zinc and retinol binding protein (RBP). Acta Derm Venereol. 1978;58(5):437-42. PMID 82355
- [Background] Dreno B, Foulc P, Reynaud A, Moyse D, Habert H, Richet H. Effect of zinc gluconate on propionibacterium acnes resistance to erythromycin in patients with inflammatory acne: in vitro and in vivo study. Eur J Dermatol. 2005 May-Jun;15(3):152-5. PMID 15908296
- [Background] Jarrousse V, Castex-Rizzi N, Khammari A, Charveron M, Dreno B. Zinc salts inhibit in vitro Toll-like receptor 2 surface expression by keratinocytes. Eur J Dermatol. 2007 Nov-Dec;17(6):492-6. doi: 10.1684/ejd.2007.0263. Epub 2007 Oct 19. PMID 17951128
- See also: Evaluation of Severity in Patients of Acne Vulgaris by Global Acne Grading System in Bangladesh — https://www.researchgate.net/publication/338964273_Evaluation_of_Severity_in_Patients_of_Acne_Vulgaris_by_Global_Acne_Grading_System_in_Bangladesh
- See also: NIH Zinc fact sheet — https://ods.od.nih.gov/factsheets/Zinc-HealthProfessional/
- See also: Drug Bank zinc gluconate — https://go.drugbank.com/drugs/DB11248
- See also: summary of zinc — https://examine.com/supplements/zinc/
- See also: Zinc for testosterone — https://supplementsinreview.com/testosterone/zinc-testosterone/
- See also: Serum Trace Elements (Zinc, Copper and Magnesium) Status in Iraqi Patients with Acne Vulgaris: (Case- Controlled Study) — https://bijps.uobaghdad.edu.iq/index.php/bijps/article/view/474
- See also: A Cross-Sectional Study on the Impact of Acne Vulgaris on the Quality of Life among High School Students in Pasig City, Philippines — http://scinet.science.ph/union/Downloads/Fil-361265_361265.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Zinc Gluconate Group: interventions: Zinc gluconate (200g/capsule) one capsule once in the morning after breakfast for 60 days.
  Adapalene 0.3% + benzoyl peroxide 2.5% gel to be applied once at night for 60 days.
  Zinc gluconate: oral zinc gluconate 200mg
  Adapalene 0.003 MG/MG / Benzoyl Peroxide 0.025 MG/MG Topical Gel [Epiduo]: Adapalene 0.3% + Benzoyl peroxide 2.5% gel applied once daily in the evening
Period: Overall Study
Arm/Group | Zinc Gluconate Group | Placebo Group
Started | 11 | 12
Completed | 8 | 8
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc Gluconate Group | Placebo Group | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  Participants
    <=18 years | 5 | 1 | 6
    Between 18 and 65 years | 3 | 7 | 10
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  Participants
    Female | 6 | 6 | 12
    Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 8 | 8 | 16
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  Participants
    Philippines | 8 | 8 | 16
Inflammatory Score [Median (Full Range); unit: units on a scale] — The inflammatory score is a grading system that measures inflammatory lesions (papules, pustules, nodules). Locations for assessment include the face, chest and back. For each location, papules, pustules and nodules are counted. A factor based on the lesion (papule=3, pustule=4, nodule=5) is multiplied to a grade equivalent to the number of lesions (0= No lesions, 1= 1-5 lesions, 2= 6-10 lesions, 3= 11-20 lesions, 4= more than 20 lesions).
  The subtotal scores are added to come up with the total inflammatory score. A maximum possible total score of 144. Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  units on a scale | 70 [43 to 110.67] | 48.5 [19.67 to 72.33] | 62.84 [19.67 to 110.67]
Global Acne Grading System score [Median (Full Range); unit: units on a scale] — The Global Acne Grading System (GAGS) is an acne severity scale. A factor is provided for each location based on size (forehead=2, right cheek=2, left cheek=2, nose=1, chin=1, chest and upper back=3). Each location is graded based on the most severe lesion present (no lesion=0, comedones=1, papules=2, pustules=3, nodules=4). The local score per location is equal to location factor multiplied by the score for the most severe lesion. The sum of local scores for all locations is the global score. Acne is rated as mild (1-18), moderate (19-30), severe (31-38), and very severe (≥39). Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
  units on a scale | 32 [25.67 to 43] | 30.33 [21 to 38.33] | 31.5 [21 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Global Acne Grading System Score
Description: changes in Global Acne Grading System (GAGS) score. Minimum score is 0, maximum score is 44. Cut off scores are as follows: no lesion (0), mild (1-18), moderate (19-30), severe (31-38), and very severe (≥39)
Time Frame: upon enrollment, at 4 weeks, at 8 weeks
Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Zinc Gluconate Group | Placebo Group
Number analyzed (Participants) | 8 | 8
score on a scale
  Initial | 32 [25.67 to 43] | 30.33 [21 to 38.33]
  4 weeks | 21.67 [19 to 29] | 27.5 [11 to 36]
  8 weeks | 14.34 [2 to 24.67] | 21.67 [7.67 to 27.67]

2. Primary Outcome: Inflammatory Score
Description: changes in inflammatory score. Minimum score is 0, maximum score is 144. Higher score indicates presence of more inflammation.
Time Frame: upon enrollment, at 4 weeks, at 8 weeks
Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Zinc Gluconate Group | Placebo Group
Number analyzed (Participants) | 8 | 8
score on a scale
  Initial | 70 [43 to 110.67] | 48.5 [19.67 to 72.33]
  4 weeks | 22.67 [12.67 to 42.38] | 47.5 [10.67 to 73.67]
  8 weeks | 8.34 [3 to 32.33] | 22.67 [10.67 to 51]

3. Secondary Outcome: Examiner's Assessment Score
Description: examiner's assessment of acne improvement graded as no improvement (0%), slight improvement (<50%), marked improvement (≥50%)
Time Frame: at 8 weeks
Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc Gluconate Group | Placebo Group
Number analyzed (Participants) | 8 | 8
Participants
  No Improvement | 0 | 0
  Slight Improvement (<50%) | 0 | 0
  Marked Improvement (≥50%) | 8 | 8

4. Secondary Outcome: Patient's Self-assessment Score
Description: patient's assessment of acne improvement graded as no improvement (0%), slight improvement (<50%), marked improvement (≥50%)
Time Frame: at 8 weeks
Population: the analysis population only consisted of participants who were able to complete 8 weeks of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Zinc Gluconate Group | Placebo Group
Number analyzed (Participants) | 8 | 8
Participants
  No improvement | 0 | 0
  Slight improvement (<50%) | 0 | 0
  Marked improvement (≥50%) | 8 | 8

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Zinc Gluconate Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc Gluconate Group (N=11) | Placebo Group (N=12)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT05096312/Prot_SAP_000.pdf